CLINICAL TRIAL: NCT02993458
Title: DASH-Sodium Trial in Adolescents
Acronym: CampDASH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: safety risks to youth in the study required early termination of the study
Sponsor: Purdue University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Johns Hopkins University (Other); Indiana University School of Medicine (Other); University of California, San Diego (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Berdine Martin, Senior Research Scientist, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01HL128834-01A1 (NIH); 1U01HL128834 (NIH)
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Blood High Pressure
Keywords: dietary patterns; blood pressure; adolescents; dietary sodium
MeSH Terms: conditions — Hypertension | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DASH diet-Low Na diet (Experimental): DASH style diet, low sodium (1500 mg/d).
  Interventions: Other: DASH diet; Other: Low Na diet
- DASH diet-High Na diet (Active Comparator): DASH style diet, high sodium (3500 mg/d).
  Interventions: Other: DASH diet; Other: High Na diet
- Usual diet-Low Na diet (Active Comparator): Diet reflecting typical dietary pattern of American adolescents, low sodium (1500 mg/d).
  Interventions: Other: Low Na diet; Other: Usual Diet
- Usual diet-High Na diet (Active Comparator): Diet reflecting typical dietary pattern of American adolescents, high sodium (3500 mg/d).
  Interventions: Other: High Na diet; Other: Usual Diet

INTERVENTIONS:
Other: DASH diet — DASH style diet rich in fruits, vegetables, and low-fat dairy foods and low in saturated fat and total fat
  Arms: DASH diet-High Na diet; DASH diet-Low Na diet
Other: Low Na diet — Sodium intake of 1500 mg/d (65 mmol, or 0.75 mg/Kcal/d), representing the Adequate Intake recommended by the Institute of Medicine.
  Arms: DASH diet-Low Na diet; Usual diet-Low Na diet
Other: High Na diet — Sodium intake of 3500 mg/d (152 mmol, or 1.73 mg/Kcal/d, representing the highest sodium intake used for adults in the DASH Sodium trial.
  Arms: DASH diet-High Na diet; Usual diet-High Na diet
Other: Usual Diet — The usual diet will include foods that provide the majority of energy for adolescents in the U.S., i.e. grain based desserts, pizza, sugary drinks,pasta, chicken, and chicken mixed dishes.
  Arms: Usual diet-High Na diet; Usual diet-Low Na diet

SUMMARY:
The Camp DASH study trial will compare the effect of two dietary patterns and two levels of sodium intake on blood pressure and blood lipids in adolescents in the upper third of distribution for blood pressure. The two dietary patterns are based on the Dietary Approaches to Stop Hypertension (DASH) trial in adults.

DETAILED DESCRIPTION:
The Camp DASH study is a controlled trial. the aim of which is to compare the effect of two dietary patterns and two levels of sodium intake on blood pressure and blood lipids in adolescents in the upper third of distribution for blood pressure. The study also assesses whether influences on blood pressure and blood lipids of dietary interventions vary according to sex, race/ethnic groups, baseline levels, and other personal characteristics. The proposed dietary interventions of DASH dietary patterns and sodium reduction have been shown to be effective in lowering blood pressure in adults. The two dietary patterns are based on the Dietary Approaches to Stop Hypertension (DASH) trial in adults. They are a Usual diet typical of what many American adolescents eat, and a DASH-type diet. The DASH diet is rich in fruits, vegetables, and low-fat dairy foods and low in saturated fat and total fat compared to the Usual diet. The two sodium levels are High reflecting current US consumption and Low reflecting current recommended intake levels. Weight will be held constant by adjusting energy intake. The study participants will live in a residence hall on the Purdue campus where all food and beverages will be provided, and meals and snacks will be supervised.

ELIGIBILITY:
Inclusion Criteria:

* White, black, Hispanic, and Asian
* SBP in the upper one-third of the distribution for their given sex, age, and height

Exclusion Criteria:

* Pre-existing lipid disorders, abnormal liver or kidney function
* Taking medications that alter mineral absorption or metabolism, affect blood pressure or lipids
* If subjects are taking dietary supplements and refuse to discontinue them 2 months prior to the study.
* Taking non-prescription illegal drugs, smoke, or drink alcohol
* Pregnancy
* Carry an epi pen for food-related allergies

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure (SBP) | End of 25 day feeding intervention
  The primary outcome is mean SBP at the end of each intervention feeding period. Mean end of intervention SBP is the average of daily readings during days 19-25 of each intervention feeding period. Blood pressure will also be measured periodically at baseline and throughout the study.
Non-HDL Cholesterol (HDLC) | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period

SECONDARY OUTCOMES:
Diastolic blood pressure (DBP) | End of 25 day feeding intervention
  The secondary outcome is mean DBP at the end of each intervention feeding period. Mean end of intervention DBP is the average of daily readings during days 19-25 of each intervention feeding period. Blood pressure will also be measured periodically at baseline and throughout the study..
Total cholesterol | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period.
HDL-cholesterol | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period
LDL-cholesterol | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period
Cholesterol:HDLC ratio | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period.
Triglycerides | End of 25 day feeding intervention
  Fasting blood samples for lipids and other variables will be drawn at the beginning and end of each feeding period
Urinary mineral excretion | End of 25 day feeding intervention
  Two 24-hr urine samples at the end of the feeding periods will be analyzed for sodium, potassium, magnesium, and calcium..
Regulators of sodium metabolism | End of 25 day feeding intervention
  Regulators of sodium homeostasis (renin, aldosterone, angiotensin) will be measured at the beginning and end of the feeding period
Augmentation index | End of 25 day feeding intervention
  Pulse wave analysis (At Cor Medical) will be used to measure changes in augmentation index (AI) with intervention to index central blood pressure.
Vasoreactivity | End of 25 day feeding intervention
  Skin flow motion (laser-doppler flowmetry) to measure diet-induced changes in vaso-reactivity will provide mechanistic information on microvascular control.

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Department of Nutrition Science, Purdue University; Berdine R Martin, PhD, Study Director — Department of Nutrition Science, Purdue University
Locations (2):
- United States (2):
  - Department of Pediatrics, IU School of Medicine, Indianapolis, Indiana
  - Department of Nutrition Science, Purdue University, West Lafayette, Indiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Chen X, Wang Y. Tracking of blood pressure from childhood to adulthood: a systematic review and meta-regression analysis. Circulation. 2008 Jun 24;117(25):3171-80. doi: 10.1161/CIRCULATIONAHA.107.730366. Epub 2008 Jun 16. PMID 18559702
- [Background] Couch SC, Saelens BE, Levin L, Dart K, Falciglia G, Daniels SR. The efficacy of a clinic-based behavioral nutrition intervention emphasizing a DASH-type diet for adolescents with elevated blood pressure. J Pediatr. 2008 Apr;152(4):494-501. doi: 10.1016/j.jpeds.2007.09.022. Epub 2007 Nov 5. PMID 18346503
- [Background] Food and Nutrition Board, Institute of Medicine. 'Sodium and chloride', Dietary Reference Intakes for Water, Potassium, Sodium, Chloride, and Sulfate. Washington, D.C.: National Academies Press; 2005. 269-423.
- [Background] Palacios C, Wigertz K, Martin BR, Braun M, Pratt JH, Peacock M, Weaver CM. Racial differences in potassium homeostasis in response to differences in dietary sodium in girls. Am J Clin Nutr. 2010 Mar;91(3):597-603. doi: 10.3945/ajcn.2009.28400. Epub 2009 Dec 9. PMID 20007307
- [Background] Palacios C, Wigertz K, Braun M, Martin BR, McCabe GP, McCabe L, Pratt JH, Peacock M, Weaver CM. Magnesium retention from metabolic-balance studies in female adolescents: impact of race, dietary salt, and calcium. Am J Clin Nutr. 2013 May;97(5):1014-9. doi: 10.3945/ajcn.112.039867. Epub 2013 Apr 3. PMID 23553157
- [Background] Palacios C, Wigertz K, Martin BR, Jackman L, Pratt JH, Peacock M, McCabe G, Weaver CM. Sodium retention in black and white female adolescents in response to salt intake. J Clin Endocrinol Metab. 2004 Apr;89(4):1858-63. doi: 10.1210/jc.2003-031446. PMID 15070956
- [Background] Rakova N, Juttner K, Dahlmann A, Schroder A, Linz P, Kopp C, Rauh M, Goller U, Beck L, Agureev A, Vassilieva G, Lenkova L, Johannes B, Wabel P, Moissl U, Vienken J, Gerzer R, Eckardt KU, Muller DN, Kirsch K, Morukov B, Luft FC, Titze J. Long-term space flight simulation reveals infradian rhythmicity in human Na(+) balance. Cell Metab. 2013 Jan 8;17(1):125-31. doi: 10.1016/j.cmet.2012.11.013. PMID 23312287
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Van Horn L, Obarzanek E, Barton BA, Stevens VJ, Kwiterovich PO Jr, Lasser NL, Robson AM, Franklin FA Jr, Lauer RM, Kimm SY, Dorgan JF, Greenlick MR. A summary of results of the Dietary Intervention Study in Children (DISC): lessons learned. Prog Cardiovasc Nurs. 2003 Winter;18(1):28-41. doi: 10.1111/j.0889-7204.2003.01007.x. PMID 12624570
- [Background] Weaver CM, Martin BR, McCabe GP, McCabe LD, Woodward M, Anderson CA, Appel LJ. Individual variation in urinary sodium excretion among adolescent girls on a fixed intake. J Hypertens. 2016 Jul;34(7):1290-7. doi: 10.1097/HJH.0000000000000960. PMID 27176144